CLINICAL TRIAL: NCT07247864
Title: A Comparative Study of Carotid Artery Stenosis Stenting With Balloon Guide Catheter Combined With Distal Filter Versus Distal Filter Alone-A Multicenter, Prospective, Open-label, Endpoint-blinded, Randomized Controlled Study
Brief Title: Balloon Guide Catheter Combined With Filter Protection for Carotid Artery Stenting
Acronym: ANGEL-BEACON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Xiaochuan Huo, Director, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KS2025109
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Carotid Artery Stenosis
Keywords: Carotid artery stenosis; Carotid Artery Stenting; Balloon Guide Catheter; Embolic Protection Device; New Ischemic Lesions
MeSH Terms: conditions — Carotid Stenosis | interventions — Embolic Protection Devices

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combined Protection Group (BGC + Filter) (Experimental): Patients in this group will undergo carotid artery stenting (CAS) using a Balloon Guide Catheter (BGC) for proximal protection combined with a distal filter protection device.
  Interventions: Device: Balloon Guide Catheter; Device: Distal Filter Protection Device
- Standard Protection Group (Filter Alone) (Active Comparator): Patients in this group will undergo carotid artery stenting (CAS) using a standard guiding catheter and a distal filter protection device alone.
  Interventions: Device: Distal Filter Protection Device

INTERVENTIONS:
Device: Balloon Guide Catheter — A catheter with a balloon at the distal tip, used to temporarily arrest flow and aspirate debris during the stenting procedure.
  Other Names: BGC
  Arms: Combined Protection Group (BGC + Filter)
Device: Distal Filter Protection Device — A mesh-type device deployed distally to the stenosis to capture embolic debris during the procedure.
  Other Names: Embolic Protection Device; EPD

SUMMARY:
This multicenter, randomized, controlled trial evaluates a combined embolic protection strategy during carotid artery stenting (CAS). Carotid artery stenosis is a major cause of stroke. While stenting is an effective treatment, the procedure itself carries a risk of dislodging plaque debris, which can travel to the brain and cause new strokes or silent brain infarctions.

Currently, a distal filter (protection device) is standardly used to catch debris. However, it may not capture all particles. This study investigates whether adding a Balloon Guide Catheter (BGC)-which temporarily stops blood flow and allows for aspiration-to the standard filter protection is more effective than using the filter alone.

Patients with symptomatic (≥50% stenosis) or asymptomatic (≥70% stenosis) carotid artery stenosis who are scheduled for stenting will be randomly assigned to one of two groups:

1. Combined Protection Group: Receiving CAS using a Balloon Guide Catheter combined with a distal filter.
2. Standard Protection Group: Receiving CAS using a distal filter alone. The primary goal is to determine if the combined approach reduces the number of new ischemic lesions detected on brain MRI within 72 hours post-procedure. The study will also assess clinical stroke events over a 90-day follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Diagnosis of extracranial carotid artery stenosis meeting one of the following criteria (measured by DSA or CTA using NASCET criteria):

   Symptomatic: TIA or non-disabling stroke in the ipsilateral carotid distribution within the past 6 months, with stenosis ≥ 50%.

   Asymptomatic: Stenosis ≥ 70%, with indication for interventional therapy.
3. Pre-treatment Modified Rankin Scale (mRS) score of 0 to 1.
4. Scheduled for carotid artery stenting (CAS) as determined by the clinical team.
5. Signed informed consent provided by the patient or their legal representative.

Exclusion Criteria:

1. Occlusion of the contralateral internal carotid artery (ICA).
2. Severe stenosis of the contralateral common carotid artery (CCA) or internal carotid artery (ICA).
3. Occlusion of the ipsilateral external carotid artery (ECA).
4. Severe stenosis of the ipsilateral intracranial segment of the internal carotid artery.
5. Severe stenosis of the vertebrobasilar artery system (excluding non-dominant vertebral artery).
6. History of previous stenting in the head or neck vessels.
7. Presence of other cerebrovascular diseases, such as intracranial aneurysms > 5 mm or vascular malformations.
8. Stroke onset within the last 7 days.
9. Pregnant or lactating women.
10. Known allergy to contrast media or stent materials (e.g., Nitinol).
11. Previous large cerebral infarction with sequelae that would interfere with the assessment of endpoint events.
12. Absolute or relative contraindications to antiplatelet therapy.
13. Clear risk of cardioembolism (e.g., atrial fibrillation, atrial flutter, intracardiac thrombus) or clear indication for anticoagulation therapy.
14. Life expectancy of less than 1 year.
15. Pre-existing neurological or psychiatric diseases that would confound neurological assessment (e.g., severe dementia).
16. Severe renal insufficiency (Glomerular Filtration Rate [GFR] < 30 ml/min).
17. Contraindications to Magnetic Resonance Imaging (MRI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of New Ischemic Lesions on Diffusion-Weighted Imaging (DWI) | Post-procedure 72 hours (plus or minus 12 hours)
  Assessed by brain MRI (DWI sequences) performed within 72 hours post-procedure. The outcome is defined as the total number of new high-signal intensity lesions observed on the post-procedural DWI compared to pre-procedural baseline (if available) or recognized as new procedural emboli.

SECONDARY OUTCOMES:
Procedural Success Rate | Intra-operative
  Defined as the successful deployment and retrieval of the stent and protection devices (Balloon Guide Catheter and/or Distal Filter) without technical failure.
Total Volume of New Ischemic Lesions on DWI | Post-procedure 72 hours (± 12 hours)
  The total volume (in milliliters) of new ischemic lesions measured on DWI MRI.
Incidence of New Symptomatic Ischemic Stroke | Post-procedure 72 hours (± 12 hours)
  Occurrence of a new ischemic stroke presenting with clinical symptoms.
Rate of Early Neurological Deterioration (NIHSS Worsening) | Post-procedure 72 hours (± 12 hours)
  Defined as an increase in the National Institutes of Health Stroke Scale (NIHSS) score of > 2 points compared to baseline.
All-Cause Mortality at 30 Days | 30 days (± 5 days)
Rate of Excellent Functional Outcome (mRS 0-1) at 30 Days | 30 days (± 5 days)
  Proportion of patients with a Modified Rankin Scale (mRS) score of 0 to 1
Rate of Functional Independence (mRS 0-2) at 30 Days | 30 days (± 5 days)
  Proportion of patients with a Modified Rankin Scale (mRS) score of 0 to 2.
Quality of Life Assessment using EuroQol Five Dimensions Questionnaire (EQ-5D-5L) at 30 Days | 30 days (± 5 days)
  The EQ-5D-5L descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels. The responses are converted into a single utility index score (ranging from less than 0 to 1, where 1 indicates full health and 0 indicates dead). Higher scores indicate better health-related quality of life.
Rate of Excellent Functional Outcome (mRS 0-1) at 90 Days | 90 days (± 7 days)
  Proportion of patients with a Modified Rankin Scale (mRS) score of 0 to 1.
Rate of Functional Independence (mRS 0-2) at 90 Days | 90 days (± 7 days)
  Proportion of patients with a Modified Rankin Scale (mRS) score of 0 to 2.
Quality of Life Assessment using EuroQol Five Dimensions Questionnaire (EQ-5D-5L) at 90 Days | 90 days (± 7 days)
  The EQ-5D-5L descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels. The responses are converted into a single utility index score (ranging from less than 0 to 1, where 1 indicates full health and 0 indicates dead). Higher scores indicate better health-related quality of life.
Incidence of Symptomatic Intracranial Hemorrhage | Post-procedure 48 hours (± 12 hours)
Incidence of Any Intracranial Hemorrhage | Post-procedure 48 hours (± 12 hours)
Incidence of Adverse Events (AEs) | Through study completion, up to 90 days
  Number of participants with adverse events.
Incidence of Serious Adverse Events (SAEs) | Through study completion, up to 90 days
  Number of participants with serious adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided